CLINICAL TRIAL: NCT02217943
Title: A Prospective, Multi-Center Study for the Evaluation of Metabolic Surgery in Subjects With Type 2 Diabetes in China
Brief Title: Prospective Metabolic Surgery in T2DM Chinese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESC-14-002
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y gastric bypass (Active Comparator): Subjects who receive a Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-Y gastric bypass
- Sleeve Gastrectomy (Active Comparator): Subjects who receive a sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass
  Arms: Roux-en-Y gastric bypass
Procedure: Sleeve gastrectomy
  Arms: Sleeve Gastrectomy

SUMMARY:
The primary goal of this study is to assess impact of metabolic surgery on glycemic control in diabetic patients.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the impact of metabolic surgery (Roux-en-Y gastric bypass [RYGB] or sleeve gastrectomy [SG]) on composite measure of glycemic control at 2 years post surgery in a Type 2 Diabetes Mellitus (T2DM) cohort of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 60 years of age (inclusive) on the date the informed consent document (ICD) is signed;
2. A body mass index (BMI) from 28 kg/m2 to 50 kg/m2 ;
3. Previously diagnosed for at least 6 months with T2DM according to World Health Organization (WHO) criteria;
4. C-peptide > 1 ng/mL (0.3 nmol/L);
5. Able and willing to comply with procedures required by the protocol; and
6. Able to comprehend and sign or, if illiterate, leave their thumb impression on the study ICD.

Exclusion Criteria:

1. History of T2DM for a duration > 10 years;
2. History of drug and/or alcohol abuse within 2 years of Screening Visit;
3. Any previous major GI surgery (e.g., any GI surgery with a resection, etc.). Previous GI surgery allowed include: appendectomy, gall bladder surgery, liver biopsies, and endoscopic procedures;
4. Scheduled concurrent surgical, non-endoscopy, procedure from Visit 1 through the end of Visit 3;
5. Women of childbearing potential who are pregnant or lactating at the time of screening, at the time of surgery, or planning to become pregnant one year or sooner after the surgery;
6. Psychiatric disorders that may affect compliance with the clinical study, including dementia, active psychosis, severe depression, or history of suicide attempts;
7. Any of the following conditions:

   1. Inflammatory diseases of the GI tract, including severe intractable esophagitis, gastric ulceration, duodenal ulceration, or specific inflammation such as Crohn's disease or ulcerative colitis that have been active within the past 10 years;
   2. End stage renal disease;
   3. Abnormal results from glutamic acid decarboxylase autoantibodies (GADA) or protein tyrosine phosphatase-like protein (IA-2A) testing; or
   4. Immunocompromised such as that resulting from chronic oral steroid use, cancer chemotherapeutic agents, or immune deficiency disorders;
8. Participation in any other clinical study (not to include registries or survey-only studies) within 30-days or 5 half-lives of an investigational drug (which ever is longer), of Visit 1 (Screening Visit) and for the duration of the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Glycemic Control - Complete Remission | 2 years
  Normal measures of glucose metabolism (glycosylated hemoglobin A1c [HbA1c] < 6% [7.0 mmol/L] and fasting plasma glucose [FPG] < 100 mg/dL [5.6 mmol/L]) for 1 year in the absence of antidiabetic medications;
Composite Measure of Glycemic Control - Partial remission | 2 years
  Hyperglycemia (HbA1c 6% - 6.4% [7.0 - 7.6 mmol/L] and FPG 100 - 125 mg/dL [5.6 mmol/L - 6.9 mmol/L]) for 1 year in the absence of anti-diabetic medications;
Composite Measure of Glycemic Control - Improvement | 2 years
  Significant reduction in HbA1c (by > 1%) or FPG (> 25 mg/dL [1.4 mmol/L]) OR reduction in HbA1c and FPG accompanied by a decrease in antidiabetic medication requirement (by discontinuing insulin or 1 oral agent, or ½ reduction in dose) for at least 1-year duration;
Composite Measure of Glycemic Control - Unchanged | 2 years
  The absence of remission or improvement as described earlier;
Composite Measure of Glycemic Control - Recurrence | 2 years
  FPG or HbA1c in the diabetic range (≥ 126 mg/dL [7.0 mmol/L] and ≥ 6.5% [7.8 mmol/L], respectively) OR need for antidiabetic medication after initial complete or partial remission.

SECONDARY OUTCOMES:
Composite Measure of Glycemic Control | 5 years
  The composite measure of glycemic control will be defined as previously described in the primary outcome measure.
Evaluation of diabetic nephropathy | 5 years
  Evaluate long-term diabetic nephropathy
Evaluation of diabetic retinopathy | 5 years
  Evaluate long-term diabetic retinopathy.
Assess changes in HbA1c | 5 years
  Assess changes in HbA1c after the procedure is performed.
Assess changes in Weight (kg) | 5 years
  Assess changes in weight after the procedure is performed.
Assess changes in BMI | 5 years
  Assess changes in BMI after the procedure is performed.
Assess changes in high-density lipoprotein (HDL) (mg/dL and mmol/L) | 5 years
  Assess changes in high-density lipoprotein (HDL) (mg/dL and mmol/L) after the procedure is performed
Assess changes in low-density lipoprotein (LDL) (mg/dL and mmol/L | 5 years
  Assess changes in low-density lipoprotein (LDL) (mg/dL and mmol/L) after the procedure is performed.
Assess changes in triglycerides (TG) (mg/dL and mmol/L) | 5 years
  Assess changes in triglycerides (TG) (mg/dL and mmol/L) after the procedure is performed.
Assess changes in cholesterol (mg/dL and mmol/L) | 5 years
  Assess changes in cholesterol (mg/dL and mmol/L) after the procedure is performed.
Assess changes in FPG (mg/dL and mmol/L) | 5 years
  Assess changes in FPG (mg/dL and mmol/L) after the procedure is performed
Assess changes in insulin (µU/mL and pmol/L) | 5 years
  Assess changes in insulin (µU/mL and pmol/L) after the procedure is performed
Assess changes in serum albumin level (g/L) | 5 years
  Assess changes in serum albumin level (g/L) after the procedure is performed
Assess changes in alanine aminotransferase (ALT) level (Unit [U]/L) | 5 years
  Assess changes in alanine aminotransferase (ALT) level (Unit [U]/L) after the procedure is performed
Assess changes in aspartate aminotransferase (AST) level (U/L) | 5 years
  Assess changes in aspartate aminotransferase (AST) level (U/L) after the procedure is performed
Assess changes in gamma-glutamyl transferase (GGT) level (U/L) | 5 years
  Assess changes in gamma-glutamyl transferase (GGT) level (U/L) after the procedure is performed
Assess changes in creatinine levels (mg/dL and mmol/L) | 5 years
  Assess changes in creatinine levels (mg/dL and mmol/L) after the procedure is performed
Assess changes in blood urea nitrogen (BUN) levels (mg/dL and mmol/L) | 5 years
  Assess changes in blood urea nitrogen (BUN) levels (mg/dL and mmol/L) after the procedure is performed
Assess changes in anti-hypertensive medication | 5 years
  Assess changes in anti-hypertensive medication after the procedure is performed
Asses the changes in lipid lowering medication | 5 years
  Asses the changes in lipid lowering medication after the procedure is performed
Assess the changes in hyperglycemia medication | 5 years
  Assess the changes in hyperglycemia medication after the procedure is performed
Assess the changes in SF-36 Health Survey | 5 years
  Assess the changes in SF-36 Health Survey after the procedure is performed

CONTACTS AND LOCATIONS:
Overall Officials: Robin Scamuffa, Study Director — Ethicon, Inc.
Locations (6):
- China (6):
  - Beijing Shijitan Hospital, Beijing
  - China-Japan Union Hospital of Jilin University, Changchun
  - Guangzhou Overseas Chinese Hospital, Guangzhou
  - Jiangsu Province Hospital, Jiangsu
  - Shanghai East Hospital, Shanghai
  - Shanghai No. 6 People's Hospital, Shanghai